CLINICAL TRIAL: NCT03453762
Title: The Effect of Lung Recruitment Maneuver on Postoperative Atelectasis in Children - Effect of Ultrasonography Guided Recruitment
Brief Title: The Effect of Lung Recruitment Maneuver on Postoperative Atelectasis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H1802-058-921
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recruitment maneuver group (Active Comparator): After anesthetic induction, recruitment maneuver is provided with positive pressure of 30 cmH2O for 10 seconds.
  Interventions: Procedure: recruitment maneuver
- Lung ultrasonography group (Experimental): After anesthetic induction, recruitment maneuver is performed, being guided by ultrasonography.
  Interventions: Procedure: ultrasonography-guided recruitment maneuver

INTERVENTIONS:
Procedure: recruitment maneuver — Recruitment maneuver is provided with positive pressure of 30 cmH2O for 10 seconds.
  Arms: Recruitment maneuver group
Procedure: ultrasonography-guided recruitment maneuver — Recruitment maneuver is guided by ultrasonography.
  Arms: Lung ultrasonography group

SUMMARY:
The investigators compare the degree of atelectasis in recovery room between conventional recruitment maneuver and ultrasonography-guided lung recruitment during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo surgery for more than 1 hour under general anesthesia
* Children under 6 years old
* American Society of Anesthesiologist Physical Status I or II

Exclusion Criteria:

* History of lung surgery
* Abnormal findings in chest x-ray
* Laparoscopic surgery
* Abdominal surgery

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative atelectasis | within 1 hour after the end of surgery
  Postoperative atelectasis is measured using lung ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Choi S, Ji SH, Jang YE, Kim EH, Kim HS, Kim JT. Effect of an ultrasound-guided lung recruitment manoeuvre on postoperative atelectasis in children: A randomised controlled trial. Eur J Anaesthesiol. 2020 Aug;37(8):719-727. doi: 10.1097/EJA.0000000000001175. PMID 32068572